CLINICAL TRIAL: NCT02893410
Title: Etude de l'Observance thérapeutique et Des Effets Secondaires Des Traitements Chez Les Patients traités Pour Polyglobulie de Vaquez et thrombocytémie Essentielle
Brief Title: Drug Observance and Side Effects of Cytoreductive Drugs in PV and ET Patients
Acronym: OUEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: OUEST (RB14.115)
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients treated with oral or sub-cutaneous drugs for polycythemia vera or essential thrombocythemia completed an unique paper questionnaire in order to describe their observance, the side effects and their own appreciation of the taken drug.

DETAILED DESCRIPTION:
During one year, all patients with PV or ET followed in our centre, and who took a drug to treat their MPN, were identified.

The investigators submitted by mail or directly at the consultation a unique questionnaire containing 25 questions concerning patients characteristics, evaluation of observance, identification of side effects and own appreciation of the drug.

After completion of the questionnaire, the patients were identified and followed to collect new data about thrombotic events or phenotypic evolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PV or ET or SMF
* Patients who took oral or sub-cutaneous drugs to treat their MPN.
* Patients who agreed to complete the questionnaire

Exclusion Criteria:

* Patients with low risk PV or ET who do not take treatment
* Patients unable to complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PV or ET who took oral or sub-cutaneous drugs to treat MPN disorders.
Sampling Method: Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Rate of adherence to drug prescription | At inclusion
  prospective evaluation in a one shot questionnaire given to each treated patient seen at the consultation distributed between december 2014 and december 2015

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Ianotto, MD, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Le Calloch R, Lacut K, Le Gall-Ianotto C, Nowak E, Abiven M, Tempescul A, Dalbies F, Eveillard JR, Ugo V, Giraudier S, Guillerm G, Lippert E, Berthou C, Ianotto JC. Non-adherence to treatment with cytoreductive and/or antithrombotic drugs is frequent and associated with an increased risk of complications in patients with polycythemia vera or essential thrombocythemia (OUEST study). Haematologica. 2018 Apr;103(4):607-613. doi: 10.3324/haematol.2017.180448. Epub 2017 Dec 15. PMID 29246923